CLINICAL TRIAL: NCT07134400
Title: Prevalence and Functional Impact of Urinary Incontinence in Women With Chronic Obstructive Pulmonary Disease Undergoing Rehabilitation: a Cross-sectional Study
Acronym: PURGE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 790-PURGE; 2025-A01834-45 (Other: ID RCB)
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Urinary Incontinence (UI); Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAD test: Patient will be ask to answer to the Leicester Cough questionnaire and the ICIQ-FLUTS questionnaire. They will also performed a PAD test.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a pathology characterized by progressive bronchial obstruction associated with an abnormal inflammatory response, leading to chronic cough, increased bronchial secretions, and irreversible destruction of alveolar walls according to the French-Language Pulmonology Society, in 2023, over 1.3 million patients were treated for this condition in France. The World Health Organization ranks COPD as the third leading cause of mortality worldwide. Historically, COPD predominantly affected men due to higher smoking rates. However, with the rise in smoking among women, recent studies have shown that the prevalence of COPD in women increased from 28 to41 perr 10,000 between 2006 and 2015. Moreover, the clinical presentation of the disease differs between genders. For equivalent smoking exposure, women appear to be more severely affected than men, experiencing greater dyspnea and a higher risk of exacerbations, leading to more frequent hospitalizations and a generally poorer quality of life.

Beyond pulmonary impairment, another clinically significant but often underestimated symptom affecting quality of life is urinary incontinence. It appears more common in individuals with COPD, particularly due to chronic cough, repeated abdominal hyperpressure, and pelvic floor muscle imbalance. A few studies have investigated the prevalence of urinary incontinence in people with COPD. One study, involving 995 individuals with COPD, suggested that 34.9% experienced urinary leakage. However, this was a subjective measure based on self-reported data via a simple questionnaire in a case-control study.

Another Swedish study estimated the prevalence of urinary incontinence in individuals with COPD at 49.6% in women and 30.3% in men, indicating that women may be at higher risk of developing this symptom. Beyond these studies, the current scientific literature remains relatively limited on this topic, while the impact on patients' quality of life appears to be significant. Among the available studies, one of the most comprehensive was published in 2013 and relied solely on self-administered questionnaires distributed to a broad population (across all disease stages) outside the rehabilitation setting.

This overlapping symptomatology-combining COPD and urinary incontinence-profoundly affects patients' quality of life, physically, psychologically, as well as socially. The consequences include limited activities, social withdrawal, diminished self-esteem, and persistent discomfort in daily interactions. This situation can lead to social anxiety or fear of leakage, resulting in absenteeism or abandonment of pulmonary rehabilitation sessions, thereby compromising the effectiveness of treatment. Reduced participation in physical activity perpetuates a vicious cycle: muscle deconditioning, sarcopenia, or even malnutrition, which worsens dyspnea, loss of autonomy, and increases the risks of frailty, infections, and hospitalizations. The study by M. A. Ramon et al. (2018) illustrates this "vicious cycle," where impaired respiratory and physical capacities are self-sustaining. Without specific screening or management strategies for urinary incontinence in this context, breaking this downward spiral and improving overall care trajectories becomes challenging.

Raising awareness about the importance of screening for stress urinary incontinence in women with COPD-particularly during pulmonary rehabilitation sessions, where these symptoms are often overlooked due to lack of knowledge and available treatments-is crucial. Such screening would enhance our understanding of the link between chronic cough, stress urinary incontinence, and quality of life. Establishing a correlation between these factors would allow for tailored care pathways and referral of certain patients to targeted pelvic floor rehabilitation.

A better understanding of this phenomenon is essential to improve functional assessment and propose adapted therapeutic approaches, which could be the subject of an interventional study in the future. This study thus represents an initial exploratory step aimed at better understanding the prevalence of urinary incontinence in women with COPD undergoing rehabilitation, as well as its impact on quality of life and cough function. It is a preliminary, observational study whose results will lay the foundation for future interventional research.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45 years or older
* Patients diagnosed with GOLD stage II to IV Chronic Obstructive Pulmonary Disease (COPD)
* Patients undergoing pulmonary rehabilitation for COPD in a specialized center
* Patients able to complete the entire pad test
* Patients with no more than 3 pregnancies in their lifetime [9]
* Patients covered by a health insurance plan
* French-speaking patients
* Patients who have not objected to participating in this research

Exclusion Criteria:

* Patients who have undergone surgery in the pelvic or thoracic region less than one year ago
* Patients under guardianship or curatorship
* Patients deprived of liberty
* Patients under legal protection (safeguarding justice)
* Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 45 suffering from COPD (stage II to IV) undergoing rehabiliation for COPD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence of urinary incontinence during rehabilitation in individuals with Chronic Obstructive Pulmonary Disease (COPD) undergoing exercise-based pulmonary rehabilitation | at enrollment
  Presence of urinary incontinence (yes/no) measured by a pad test ≥ 1 gram at the end of the session

SECONDARY OUTCOMES:
severity of urinary incontinence (if detected) | at enrollment
  Weigh of the pad test in gram. , an increase of 1 to 10 g represents mild incontinence, 11 to 50 g represents moderate incontinence and > 50 g represents severe incontinence.
Impact of urinary incontinence on quality of life | at enrollement
  score at the ICIQ FLUTS
Impact of chronic cough on quality of life | at enrollement
  scored with the Leicester Couch Questionnaire
relation between cough severity and urinary incontinence | at enrollement
  correlation between Leicester Cough questionnaire and ICIQ FLUTS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christophe ROMANET, Principal Investigator — Hôpital Paris Saint Joseph
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No